CLINICAL TRIAL: NCT04958031
Title: A Randomized, Double-Blind, Placebo-Controlled Trial To Evaluate the Safety, Tolerability, and Pharmacodynamics of CVL-871 in Subjects With Dementia-Related Apathy
Brief Title: A Trial of the Safety, Tolerability, and Pharmacodynamics of CVL-871 in Subjects With Dementia-Related Apathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVL-871-2001; IND 150,086 (Other: IND)
Record Dates: First submitted 2021-06-08; First posted 2021-07-12 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Apathy in Dementia
Keywords: Dementia; Apathy
MeSH Terms: conditions — Dementia; Lethargy

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator
Masking Description: • Double Blind: two or more parties are unaware of the intervention assignment (Blinded: Participant, Caregiver, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CVL-871 1.0 mg (Experimental): Participants will receive CVL-871 tablets orally QD up to the maximum dose of 1.0 milligrams (mg) until Day 85 during the treatment period.
  Interventions: Drug: CVL-871 1.0 mg
- CVL-871 3.0 mg (Experimental): Participants will receive CVL-871 tablets orally QD up to the maximum dose of 3.0 milligrams (mg) until Day 85 during the treatment period.
  Interventions: Drug: CVL-871 3.0 mg
- Placebo (Placebo Comparator): Participants will receive a placebo matched to CVL-871 tablets orally QD until Day 85 during the treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CVL-871 1.0 mg — CVL-871 1.0 mg, oral (tablet), once per day for 12 weeks (stepped up-titration of dose days 1-7)
  Arms: CVL-871 1.0 mg
Drug: CVL-871 3.0 mg — CVL-871 3.0 mg QD oral (tablet), once per day for 12 weeks (stepped up-titration of dose days 1-21)
  Arms: CVL-871 3.0 mg
Drug: Placebo — Placebo QD, oral (tablet), once per day for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether CVL-871 is safe and tolerable in patients with Dementia-Related Apathy and if CVL-871 shows changes in clinical measurements of apathy.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for apathy in neurocognitive disorders
* Clinically significant apathy
* Mild to Moderate Dementia (AD, FTD, VAD, or DLB)

Exclusion Criteria:

* Other significant psychiatric disorder(s)
* Other neurological disorders (other than AD, FTD, VAD, or DLB)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Treatment Emergent Adverse Events (TEAEs) | From first dose of study drug up to Week 16 (follow-up period)
  Any AE occurring following the start of treatment or occurring before treatment but increasing in severity afterward were counted as treatment-emergent AE (TEAE)
Incidence of clinically significant changes in electrocardiogram (ECG) results | Baseline up to Week 16 or early termination (ET)
  Assessment of clinically significant changes in QT intervals measured by 12-lead ECG recording after the participant has been supine and at rest for at least 5 minutes
Incidence of clinically significant changes in clinical laboratory results | Baseline up to Week 14 or early termination (ET)
Incidence in clinically significant changes in vital sign measurements | Baseline up to Week 14 or early termination (ET)
  Assessment of clinically significant changes in vital signs including temperature, systolic and diastolic blood pressure, and heart rate.
Incidence of clinically significant changes in physical and neurological examination results | Screening up to Week 16 or early termination (ET)
Clinically significant findings in suicidality assessed using the Columbia Suicide-Severity Rating Scale (C-SSRS) | Baseline up to Week 14 (follow up period)
  The C-SSRS rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent).

SECONDARY OUTCOMES:
Change from baseline in the Dementia Apathy Interview and Rating (DAIR) score | Baseline up to Week 12 or early termination (ET)
  The Dementia Apathy Interview Rating (DAIR) is a 16-item structured interview with the primary caregiver designed to assess illness-related changes in motivation, emotional responsiveness, and engagement. The total apathy score is a sum of all items reflecting change (items for which there is no change are not rated), divided by the number of items completed, with higher scores representing greater average apathy. In addition, the frequency of these behaviors is assessed; higher scores represent more frequent apathy-related behavior.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (19):
- United States (16):
  - Scottsdale, Arizona, Scottsdale, Arizona
  - Little Rock, Arkansas, Little Rock, Arkansas
  - San Diego, California, San Diego, California
  - Santa Ana, California, Santa Ana, California
  - New Haven, Connecticut, New Haven, Connecticut
  - Delray Beach, Florida, Delray Beach, Florida
  - Miami, Florida, Miami, Florida
  - Orlando, Florida, Orlando, Florida
  - Wellington, Florida, Wellington, Florida
  - Decatur, Georgia, Decatur, Georgia
  - Plymouth, Massachusetts, Plymouth, Massachusetts
  - Staten Island, New York, Staten Island, New York
  - Columbus, Ohio, Columbus, Ohio
  - Abington, Pennsylvania, Abington, Pennsylvania
  - Charleston, South Carolina, Charleston, South Carolina
  - Fairfax, Virginia, Fairfax, Virginia
- Canada (3):
  - Calgary, Alberta, Calgary, Alberta
  - Victoria, British Columbia, Victoria, British Columbia
  - Toronto, Ontario, Toronto, Ontario